CLINICAL TRIAL: NCT04924517
Title: The Effect of 4 Days of Extended Evening Fasting on Metabolic Health, Energy Balance and Appetite
Brief Title: Extended Evening Fasting: Metabolic Health and Energy Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham Trent University (Other)
Responsible Party: Principal Investigator, William Mode, Principle Investigator, Nottingham Trent University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WM_EEF_2021
Record Dates: First submitted 2021-05-24; First posted 2021-06-14 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Chrononutrition; Energy balance; Intermittent fasting; Appetite hormones
MeSH Terms: conditions — Obesity; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake two conditions in a randomised order with at least four weeks in between trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Evening Fasting (Experimental): Participants will eat between 8am-4pm
  Interventions: Behavioral: Extended Evening Fasting
- Control (Active Comparator): Participants will eat between 8am-8pm
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Extended Evening Fasting — Participants will undertake 4 days of extended evening fasting (feeding between 8am-4pm). The participants will visit the laboratory on day 1, following a 16 h fast, where baseline measures will be taken and the response to a standardised meal will take place. The participant will also have an opportunity to feed ad-libitum before they leave the laboratory. The participant will continue to adhere to the feeding window on day 2 and day 3, although this will be in free-living conditions. On day 4, the participant will arrive back to the lab for post-intervention assessment, identical in format to day 1 with a metabolic assessment and energy intake assessment via a ad-libitum meal.
  Arms: Extended Evening Fasting
Behavioral: Control — Participants will undertake 4 days of a standard western feeding pattern (feeding between 8am-8pm). The participants will visit the laboratory on day 1, following a 12 h fast, where baseline measures will be taken and the response to a standardised meal will take place. The participant will also have an opportunity to feed ad-libitum before they leave the laboratory. The participant will continue to adhere to the feeding window on day 2 and day 3, although this will be in free-living conditions. On day 4, the participant will arrive back to the lab for post-intervention assessment, identical in format to day 1 with a metabolic assessment and energy intake assessment via a ad-libitum meal.
  Arms: Control

SUMMARY:
This study will compare metabolic and feeding behaviour responses to 4 days of extended evening fasting vs. a control trial

DETAILED DESCRIPTION:
Humans have evolved as a diurnal species, internally governed by the circadian system, which dictates our hormone regulation. 'Chrononutrition' is a sub-discipline which combines food timing with circadian physiology. The most popular method of time-restricted feeding in the UK is to skip breakfast. However, data from several meta-analysis have shown that skipping breakfast is associated with weight gain and insulin resistance, likely due to eating later into the evening/night and therefore, out of sync with our circadian rhythm. Recent research has shown that skipping dinner (evening fasting) has improved markers of cardio-metabolic health in clinical populations, although these are typically from longer-term studies. Despite these promising findings, it is not yet known whether these findings are population specific.

Therefore, the investigators are interested in examining the metabolic response pre and post intervention to see whether these promising findings can translate into a healthy population. Furthermore, the investigators will be monitoring subjective appetite, energy intake and expenditure to assess whether there is any short-term adaptation to a specific feeding window.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers.

  * Have maintained a stable weight for 6 months (self-reported).
  * No history of gastric, digestive, cardiovascular or renal disease (self reported).
  * Female specific: must be using a monophasic, low dose combined OCP (containing less than 50μg oestradiol and a synthetic progestin) OR females with regular menstrual cycles (self-reported).

Exclusion Criteria:

* Severe food allergies, dislike or intolerance of study foods or drinks.

  * Currently undergoing a lifestyle intervention (structured diet or exercise)
  * Diagnosis of a condition or currently undergoing treatment therapy known to affect glucose or lipid metabolism (e.g., type-2 diabetes, taking statins), or contraindications to exercise.
  * Use of medication or supplements that may affect hormone concentrations.
  * Excessive alcohol consumption (>14 units/week).
  * Intensive training schedule (>10 hours/week).
  * Female specific: currently pregnant or breastfeeding, the use of any hormonal contraception, and the self-reporting of short (<24 d), long (>35 d), or irregular menstrual cycles.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-06-14 (Estimated); Study Completion 2022-06-14 (Estimated)

PRIMARY OUTCOMES:
Glycaemic control (Baseline) | 3.5 hours following the standardised breakfast meal on day 1.
  A metabolic assessment lasting 3.5 hours will take place following a standardised, laboratory-based meal. The investigators will be taking periodic capillary and venous blood samples to measure post-prandial glucose and insulin, which together comprise 'glycaemic control'.
Glycaemic control (Post intervention) | 3.5 hours following the standardised breakfast meal on day 4.
  A metabolic assessment lasting 3.5 hours will take place following a standardised, laboratory-based meal. The investigators will be taking periodic capillary and venous blood samples to measure post-prandial glucose and insulin, which together comprise 'glycaemic control'.
Energy Intake (Kilocalories) | Day 1 to day 4.
  Energy intake will be measured both during lab and outside of the laboratory when the participants are free-living. During lab, energy intake will be measured through ad-libitum feeding buffet where 20 minutes will be permitted to eat as much or as little as they desire, until 'comfortably full and satisfied', followed by post-feeding measurement of the remaining food. Outside of laboratory feeding will also be monitored through food diary's and weighing any investigator issued meals.
Energy expenditure | Day 1 to day 4.
  Energy expenditure will be measured via a chest-worn device (Actiheart) which combines heart rate and accelerometry to gauge calories expended.

SECONDARY OUTCOMES:
Cortisol awakening response | Five samples will be collected by the participant within the first hour of waking on day 5.
  The cortisol awakening response will be measured on the final morning of each trial.
Visual Analogue Scale for Subjective Ratings of Appetite | Every 2 hours between 8am-10pm from day 1 to day 4.
  Subjective appetite will be measured on mobile devices via a software which replicates a 100mm visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, desire to eat and prospective food consumption.
  (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Acylated Ghrelin (appetite hormone) | 3.5 hours following the standardised breakfast meal on day 1 and day 4.
  Acylated Ghrelin will be measured from the venous samples taken during the post-prandial period following the standardised meal.
PYY (appetite hormone) | 3.5 hours following the standardised breakfast meal on day 1 and day 4.
  PYY will be measured from the venous samples taken during the post-prandial period following the standardised meal.
Carbohydrate oxidation | During laboratory visits on day 1 and day 4 [baseline, 60min, 120min, 180min]
  Investigators will be collecting expired air into Douglas bags, and measuring the VO2 and VCO2 concentration to calculate carbohydrate oxidation.
Fat oxidation | During laboratory visits on day 1 and day 4 [baseline, 60min, 120min, 180min]
  Investigators will be collecting expired air into Douglas bags, and measuring the VO2 and VCO2 concentration to calculate fat oxidation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Nottingham, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Background] Ravussin E, Beyl RA, Poggiogalle E, Hsia DS, Peterson CM. Early Time-Restricted Feeding Reduces Appetite and Increases Fat Oxidation But Does Not Affect Energy Expenditure in Humans. Obesity (Silver Spring). 2019 Aug;27(8):1244-1254. doi: 10.1002/oby.22518. PMID 31339000
- [Background] Hutchison AT, Regmi P, Manoogian ENC, Fleischer JG, Wittert GA, Panda S, Heilbronn LK. Time-Restricted Feeding Improves Glucose Tolerance in Men at Risk for Type 2 Diabetes: A Randomized Crossover Trial. Obesity (Silver Spring). 2019 May;27(5):724-732. doi: 10.1002/oby.22449. Epub 2019 Apr 19. PMID 31002478
- [Background] Templeman I, Gonzalez JT, Thompson D, Betts JA. The role of intermittent fasting and meal timing in weight management and metabolic health. Proc Nutr Soc. 2020 Feb;79(1):76-87. doi: 10.1017/S0029665119000636. Epub 2019 Apr 26. PMID 31023390
- [Background] Popkin BM. The nutrition transition and obesity in the developing world. J Nutr. 2001 Mar;131(3):871S-873S. doi: 10.1093/jn/131.3.871S. PMID 11238777
- [Background] Allison KC, Goel N. Timing of eating in adults across the weight spectrum: Metabolic factors and potential circadian mechanisms. Physiol Behav. 2018 Aug 1;192:158-166. doi: 10.1016/j.physbeh.2018.02.047. Epub 2018 Feb 24. PMID 29486170
- [Background] St-Onge MP, Ard J, Baskin ML, Chiuve SE, Johnson HM, Kris-Etherton P, Varady K; American Heart Association Obesity Committee of the Council on Lifestyle and Cardiometabolic Health; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; and Stroke Council. Meal Timing and Frequency: Implications for Cardiovascular Disease Prevention: A Scientific Statement From the American Heart Association. Circulation. 2017 Feb 28;135(9):e96-e121. doi: 10.1161/CIR.0000000000000476. Epub 2017 Jan 30. PMID 28137935